CLINICAL TRIAL: NCT04245189
Title: EUS Based Prevalence of Chronic Pancreatitis in Alcoholic Cirrhosis: Any Difference Between Alcoholic and Non-alcoholic Patients
Brief Title: EUS Based Prevalence of Chronic Pancreatitis in Alcoholic Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: AIG-G-EUSCP
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Alcoholic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Endoscopic ultrasound for detection of Chronic pancreatitis — Presence of Chronic pancreatitis in alcoholic cirrhosis patients.

SUMMARY:
Alcohol is the common precipitating factor for both cirrhosis of liver as well as alcohol related chronic pancreatitis. However, in real life clinical setting, clinicians do not frequently see many cases of symptomatic pancreatitis in patients who present with features of cirrhosis of liver. On the contrary, in some patients presenting with alcohol related chronic pancreatitis, evidence of cirrhosis of liver is observed on imaging without other clinical features of cirrhosis.

DETAILED DESCRIPTION:
The data on exact incidence of chronic pancreatitis in patients with alcoholic cirrhosis is scarce and there are no data to support or refute as to whether the incidence is same between alcoholic cirrhosis or cirrhosis due to any other cause. The co-existence of cirrhosis and chronic pancreatitis in alcoholics vary between 0.04 - 6%.

However, till now no study has been conducted to evaluate the incidence of CP in patients with alcoholic cirrhosis of liver. In this study, the investigators propose to assess the incidence of chronic pancreatitis in patients of ethanol related cirrhosis of liver and compare the same with patients of cryptogenic liver cirrhosis and hepatitis B and C related liver cirrhosis. This would be one of the few studies till date, to use EUS as the diagnostic modality.

The patients of cirrhosis would be categorized based on their Child Pugh criteria into three categories. All these patients would undergo EUS at the Institute and chronic pancreatitis screening would be considered positive if they fulfill the Rosemont criteria for chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

• Patients with diagnosis of ethanol related cirrhosis of liver who complains of central abdominal pain without any other identifiable cause of pain would be enrolled in the study.

Exclusion Criteria:

* Any patients with evidence of Hepatocellular carcinoma , autoimmune hepatitis related CLD, and PBC would be excluded.
* Patients any co-existent other malignancy, sepsis, pregnancy.
* An informed consent would be signed by the patient and any patient not willing to be a part of the study will be excluded.

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients attending the Hepatology unit of AIG Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pancreatitis in alcoholic cirrhotics as per Rosemont criteria . | 3 days
  To assess the incidence of chronic pancreatitis in patients of ethanol related cirrhosis of liver and compare the same with patients of cryptogenic liver cirrhosis, hepatitis B and C related liver cirrhosis.

SECONDARY OUTCOMES:
Assessment of Pain. | 3 days
  Visual Analogue Scale (VAS) measures pain intensity based on observer assessment on a scale from 1 to 10, where higher values indicate more intense pain.
Pancreatic duct size. | 3 days
  In patients found to have Chronic pancreatitis -Pancreatic duct size would be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Mithun Sharma, Principal Investigator — AIG Hospitals
Locations (1):
- Asian Institute of Gastroenterology Hospitals, Hyderabad, Telangana, India

REFERENCES:
- [Background] Stevens T, Parsi MA. Endoscopic ultrasound for the diagnosis of chronic pancreatitis. World J Gastroenterol. 2010 Jun 21;16(23):2841-50. doi: 10.3748/wjg.v16.i23.2841. PMID 20556829
- [Background] Catalano MF, Sahai A, Levy M, Romagnuolo J, Wiersema M, Brugge W, Freeman M, Yamao K, Canto M, Hernandez LV. EUS-based criteria for the diagnosis of chronic pancreatitis: the Rosemont classification. Gastrointest Endosc. 2009 Jun;69(7):1251-61. doi: 10.1016/j.gie.2008.07.043. Epub 2009 Feb 24. PMID 19243769
- [Background] Aparisi L, Sabater L, Del-Olmo J, Sastre J, Serra MA, Campello R, Bautista D, Wassel A, Rodrigo JM. Does an association exist between chronic pancreatitis and liver cirrhosis in alcoholic subjects? World J Gastroenterol. 2008 Oct 28;14(40):6171-9. doi: 10.3748/wjg.14.6171. PMID 18985807